CLINICAL TRIAL: NCT02694094
Title: Impact of Ketogenic Diets on Cardiovascular Health in Adults With Epilepsy
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00070557
Record Dates: First submitted 2016-02-16; First posted 2016-02-29 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia; Carotid Intimal Medial Thickness 1; Seizure; Epilepsy; Cardiovascular Disease; Cerebrovascular Disease; Heart Disease; Coronary Disease
Keywords: cholesterol; seizure; epilepsy; ketogenic; diet
MeSH Terms: conditions — Hypercholesterolemia; Carotid Intimal Medial Thickness 1; Seizures; Epilepsy; Cardiovascular Diseases; Cerebrovascular Disorders; Heart Diseases; Coronary Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults on Chronic ketogenic diets: Adults who have been on Modified Atkins or ketogenic diets for over 1 year
  Interventions: Dietary Supplement: Modified Atkins or Ketogenic Diet
- Adults naive to ketogenic diets: Adults who have never been on Modified Atkins or ketogenic diets

INTERVENTIONS:
Dietary Supplement: Modified Atkins or Ketogenic Diet — Biochemical and vascular parameters will be compared from adults who have been on ketogenic diet therapy for > 12 months to adults naive to ketogenic diet therapy. In addition, adults naive to diet therapy who subsequently begin diet therapy will have these same parameters followed over time.
  Groups: Adults on Chronic ketogenic diets

SUMMARY:
This research is being done to evaluate the short term and long term effects of ketogenic diets on measures of cardiovascular health. Such measures include cholesterol levels, blood pressure, weight, and thickening of the blood vessel wall over time. Adults aged 18 or older who are already on a ketogenic diet for at least 12 months or who are interested in beginning on the modified Atkins diet may join.

DETAILED DESCRIPTION:
If participants agree to be in this study, the investigators will ask the participants to do the following things:

At Initial enrollment for both longterm ketogenic diet and new modified Atkins diet participants

* Review of calendars (showing seizures) and 3-day food record
* Check height and weight, blood pressure, skin-fold thickness and waist circumference
* Standard modified Atkins diet clinic labs will be drawn as well as levels of low density lipoprotein (LDL) fractions, fatty acids, and apolipoproteins B and A-1
* Participant will receive a high-resolution ultrasound of the carotid arteries in the neck performed either the day of enrollment or within 1 month of enrollment

At follow-up clinic visits (month 3 and month 6) for new modified Atkins diet participants

* Review of calendars and food records
* Labs repeated - standard modified Atkins diet clinic labs as well as levels of low density lipoprotein (LDL) fractions, fatty acids, and apolipoproteins B and A-1
* Check height and weight, blood pressure, skin-fold thickness and waist circumference

At follow-up clinic visits (month 12 and month 24) for new modified Atkins diet participants

* Review of calendars and food records
* Labs repeated - standard modified Atkins diet clinic labs as well as levels of low density lipoprotein (LDL) fractions, fatty acids, and apolipoproteins B and A-1
* Check height and weight, blood pressure, skin-fold thickness and waist circumference
* Participants will receive a high-resolution ultrasound of the carotid arteries in the neck performed either the day of follow-up or within 1 month of follow-up

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body mass index (BMI) > 18.5
* Stable antiepileptic drug regimen for > 1 month.

Exclusion Criteria:

* < 18 years of age
* Body mass index (BMI) < 18.5
* Changes in antiepileptic drug regimen < 1 month prior to participation
* Previous cardiovascular event or treatment ((including myocardial infarction, stroke, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI))
* Acute pancreatitis
* Unwilling to restrict carbohydrates
* Kidney disease
* Contraindicated metabolic or mitochondrial disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be drawn from among participants in the Johns Hopkins Adult Epilepsy Diet Center and Johns Hopkins Epilepsy Center who are age 18 or older, with body mass index (BMI) > 18.5, and on a stable antiepileptic drug regimen for > 1 month.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2016-03; Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in carotid artery intima-media thickness (mm) measured by carotid artery ultrasound | Baseline and 12 months post diet implementation
  Carotid artery ultrasound will be used to measure the change in average intima-media thickness over time with comparisons between baseline and 12 months of diet therapy.
Change in LDL fractions (nmol/L) | Baseline and 12 months post diet implementation
  The change in levels of fasting serum low density lipoprotein (LDL) fractions (nmol/L) will be measured over time with comparisons between baseline and 12 months of diet therapy.

SECONDARY OUTCOMES:
Change in LDL fractions (nmol/L) | Baseline and 3 months post diet implementation
  The change in levels of fasting serum low density lipoprotein (LDL) fractions (nmol/L) will be measured over time with comparisons between baseline and 3 months of diet therapy.
Change in apolipoproteins (mg/dL) | Baseline and 3 months post diet implementation
  The change in fasting serum levels of apolipoproteins B and A-1 will be measured over time with comparisons between baseline and 3 months of diet therapy.
Change in apolipoproteins (mg/dL) | Baseline and 6 months post diet implementation
  The change in fasting serum levels of apolipoproteins B and A-1 will be measured over time with comparisons between baseline and 6 months of diet therapy.
Change in apolipoproteins (mg/dL) | Baseline and 12 months post diet implementation
  The change in fasting serum levels of apolipoproteins B and A-1 will be measured over time with comparisons between baseline and 12 months of diet therapy.
Change in apolipoproteins (mg/dL) | Baseline and 24 months post diet implementation
  The change in fasting serum levels of apolipoproteins B and A-1 will be measured over time with comparisons between baseline and 24 months of diet therapy.
Change in LDL fractions (nmol/L) | Baseline and 6 months post diet implementation
  The change in levels of fasting serum low density lipoprotein (LDL) fractions (nmol/L) will be measured over time with comparisons between baseline and 6 months of diet therapy.
Change in LDL fractions (nmol/L) | Baseline and 24 months post diet implementation
  The change in levels of fasting serum low density lipoprotein (LDL) fractions (nmol/L) will be measured over time with comparisons between baseline and 24 months of diet therapy.
Change in carotid artery intima-media thickness (mm) measured by carotid artery | Baseline and 24 months post diet implementation
  Carotid artery ultrasound will be used to measure the change in average intima-media thickness over time with comparisons between baseline and 24 months of diet therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie C Cervenka, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald TJW, Diaz-Arias L, Vizthum D, Henry-Barron BJ, Schlechter H, Kossoff EH, Cervenka MC. Six-month effects of modified Atkins diet implementation on indices of cardiovascular disease risk in adults with epilepsy. Nutr Neurosci. 2022 Jul;25(7):1548-1557. doi: 10.1080/1028415X.2021.1875301. Epub 2021 Jan 23. PMID 33487129
- See also: Ketogenic Diet Therapy for Epilepsy — https://www.hopkinsmedicine.org/neurology_neurosurgery/centers_clinics/epilepsy/diet-therapy.html